CLINICAL TRIAL: NCT04086121
Title: An Open Label Extension Study to Assess the Long Term Safety of Treatment With BI 655130 Administered Subcutaneously in Adult Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Test the Long-term Safety of BI 655130 in Patients With Atopic Eczema Who Took Part in Study 1368-0032
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1368-0037
Record Dates: First submitted 2019-09-10; First posted 2019-09-11 (Actual); Results first posted 2022-05-18 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — spesolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Spesolimab 600 mg (Experimental): 600 milligrams (mg) solution for subcutaneous (SC) injection of BI 655130 (Spesolimab) were to administered subcutaneously every 4 weeks.
  All patients will return 16 weeks post the last treatment for an End of Study (EOS) visit.
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — Solution for SC injection
  Other Names: BI 655130

SUMMARY:
To assess the long term safety and efficacy of treatment with BI 655130 in patients with AD who have completed and have responded to treatment in the parent study 1368-0032

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent in accordance with Good Clinical Practice (GCP) and local legislation prior to the start of any screening procedures
* Patients who completed the 1368-0032 trial and did not prematurely discontinue treatment prior to week 16, and; In the 1368-0032 re-allocation period (V7 to V11):

  * If an original non-responder from week 16 (V7), attained at least EASI 50 by last infusion (week 28) or by the EOS.
  * If an original responder from week 16 (V7) completed the last visit Week 28 (EOS) or dropped to a EASI 50 score prior to Week 28.
* Women of childbearing potential (WOCBP)1 must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly for the duration of the trial and 16 weeks after last study drug administration. A list of contraception methods meeting these criteria is provided in the patient information.

Exclusion Criteria:

* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Any new documented active or suspected malignancy except appropriately treated basal cell carcinoma, squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Use of any restricted medication: or any drug considered likely to interfere with the safe conduct of the study, as assessed by the investigator.
* Active systemic infections during the last two weeks prior to first drug administration.
* Currently enrolled in another investigational device or drug trial, except for 1368-0032.
* Any condition which would prevent the patient continuing on treatment in this trial 1368-0037
* Evidence of a current or previous disease, medical condition (including chronic alcohol or drug abuse or any condition) other than AD, surgical procedure, psychiatric or social problems, medical examination finding (including vital signs and ECG), or laboratory value at the screening outside the reference range that in the opinion of the investigator is clinically significant and would make the study participant unreliable to adhere to the protocol, comply with all study visits/procedures or to complete the trial, compromise the safety of the patient or compromise the quality of the data.
* History of allergy/hypersensitivity to the systemically administered trial medication agent or its excipients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (7):
  - CCT Research, Scottsdale, Arizona
  - Clinical Physiology Associates, Fort Myers, Florida
  - Finlay Medical Research Corp, Miami, Florida
  - ForCare Clinical Research, Inc., Tampa, Florida
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Dermatology Treatment and Research Center, PA, Dallas, Texas
- Innovaderm Research Inc., Montreal, Quebec, Canada
- Japan (2):
  - Tennocho Ekimae Dermatology and Allergology, Kanagawa, Yokohama
  - Tokyo Medical University Hachioji Medical Center, Tokyo, Hachioji

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open label extension clinical trial was planned to offer all patients who completed the clinical trial 1368-0032 (NCT03822832) as planned, the option to continue to receive BI 655130 treatment if they have responded to treatment and meet all criteria for study entry.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Spesolimab 600 mg
Started | 14
Completed | 0
Not Completed | 14
Not completed — Other than listed | 8
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): This patient set includes all randomized patients who received at least one dose of study drug.
Arm/Group | Spesolimab 600 mg
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.2 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Emergent Adverse Events (AEs) at Week 48
Description: Number of patients with treatment emergent adverse events (AEs) at week 48. The treatment emergent adverse event refer to the adverse event with an onset between start of treatment and end of the 16-week residual effect period after the last dose of trial medication.
Time Frame: From first dose until Week 48, up to 48 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Spesolimab 600 mg
Number analyzed (Participants) | 14
Participants | 9

2. Secondary Outcome: Percentage Change From Baseline in the Eczema Area and Severity Index (EASI) Score at Week 48
Description: The EASI scoring system is used routinely in patients with psoriasis to describe signs and severity of the disease. It assesses the extent of disease at four body sites and measures four clinical signs: erythema, induration/papulation, excoriation, and lichenification (each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe)). The EASI score was obtained by weight-averaging these 4 scores, resulting in the EASI score ranges from 0 (clear) to 72 (very severe), with higher score indicating more severe disease extent and clinical signs. The percent change from baseline in EASI is calculated as: (EASI at week 48 - EASI at baseline) / EASI at baseline * 100%.
Time Frame: At baseline and at Week 48.
Population: Full analysis set (FAS): This patient set includes all patients in the SAF who had a baseline measurement and at least one post-baseline measurement for the secondary endpoint, Eczema Area and Severity Index (EASI) Total Score.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Spesolimab 600 mg: 600 milligrams (mg) solution for subcutaneous (SC) injection of BI 655130 (Spesolimab) were to administered subcutaneously every 4 weeks, up to 4 years (204 weeks) of End of Treatment (EOT).
  All patients will return 16 weeks post the last treatment for an End of Study (EOS) visit.
Arm/Group | Spesolimab 600 mg
Number analyzed (Participants) | 9
Percent change | -3.74 (81.99)

3. Secondary Outcome: Percentage of Patients With a 50% Improvement From Baseline in EASI (EASI50) at Week 48
Description: The EASI scoring system is used routinely in patients with psoriasis to describe signs and severity of the disease. It assesses the extent of disease at four body sites and measures four clinical signs: erythema, induration/papulation, excoriation, and lichenification (each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe)). The EASI score was obtained by weight-averaging these 4 scores, resulting in the EASI score ranges from 0 (clear) to 72 (very severe), with higher score indicating more severe disease extent and clinical signs. [(EASI at week 48 - EASI at baseline) / EASI at baseline * 100%] ≥ 50%, then EASI50 = 1.
Time Frame: At baseline and at Week 48.
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Spesolimab 600 mg
Number analyzed (Participants) | 9
Percentage of participants | 33.3

4. Secondary Outcome: Percentage of Patients With a 75% Improvement From Baseline in EASI (EASI75) at Week 48
Description: The EASI scoring system is used routinely in patients with psoriasis to describe signs and severity of the disease. It assesses the extent of disease at four body sites and measures four clinical signs: erythema, induration/papulation, excoriation, and lichenification (each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe)). The EASI score was obtained by weight-averaging these 4 scores, resulting in the EASI score ranges from 0 (clear) to 72 (very severe), with higher score indicating more severe disease extent and clinical signs. [(EASI at week 48 - EASI at baseline) / EASI at baseline * 100%] ≥ 75%, then EASI75 = 1.
Time Frame: At baseline and at Week 48.
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Spesolimab 600 mg
Number analyzed (Participants) | 9
Percentage of participants | 22.2

5. Secondary Outcome: Change From Baseline in SCORing of Atopic Dermatitis (SCORAD) at Week 48
Description: The SCORing of Atopic Dermatitis (SCORAD) index assesses elements: extent of disease, disease severity and subjective symptoms. The SCORAD consists of three elements: extent of disease, intensity of disease, and subjective symptoms (Pruritus and Sleep Loss). These 3 aspects: extent of disease (A: score range 0-1-2), disease severity (B: score range 0-18), and subjective symptoms (C: score range 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103 for SCORAD score. The SCORAD range from 0 (no disease) to 103 (severe disease). The higher the SCORAD score, the more severe the Atopic Dermatitis is.
Time Frame: At baseline and at Week 48.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Spesolimab 600 mg
Number analyzed (Participants) | 9
Score on a scale | -10.07 (66.04)

6. Secondary Outcome: Percentage of Patients Achieving at Least a 2-grade Reduction From Baseline to Clear (0) or Almost Clear (1) in Investigator Global Assessment (IGA) at Week 48
Description: The IGA scale allows investigators to assess overall disease severity at one given time point, and it consists of a five-point severity scale from clear to very severe disease (0= clear,1 =almost clear, 2 = mild disease, 3 = moderate disease, 4= severe disease). The IGA scale uses clinical characteristics of erythema, infiltration, papulation, oozing and crusting as guidelines for the overall severity assessment.
Time Frame: At baseline and at Week 48.
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Spesolimab 600 mg
Number analyzed (Participants) | 9
Percentage of participants | 22.2

ADVERSE EVENTS:
Time Frame: From first dose until last dose + 16 weeks, up to 765 days.
Description: Safety analysis set (SAF): This patient set includes all randomized patients who received at least one dose of study drug.
Arm/Group | Spesolimab 600 mg
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimab 600 mg (N=14)
COVID-19 pneumonia (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimab 600 mg (N=14)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Asymptomatic COVID-19 (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 3
Skin infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Tinea versicolour (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Upper respiratory tract infection bacterial (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Splinter (Injury, poisoning and procedural complications) | 1
Vitamin B12 decreased (Investigations) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Cervical radiculopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to sponsor decision. The planned treatment period of 4 years was not reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT04086121/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT04086121/SAP_001.pdf